CLINICAL TRIAL: NCT01564290
Title: Use of Probiotic Yogurt in the Treatment of Acute Diarrhea in Children: A Randomized Double-blind Trial
Brief Title: Use of Probiotic Yogurt in the Treatment of Acute Diarrhea in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro Pediatrico Albina de Patino (Other)
Responsible Party: Principal Investigator, Carlos Teran, Teaching and Research chief, Centro Pediatrico Albina de Patino
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: protprobiot2010
Record Dates: First submitted 2011-10-29; First posted 2012-03-27 (Estimated); Last update posted 2012-03-27 (Estimated); Status verified 2012-03

CONDITIONS: Acute Diarrhea; Acute Gastroenteritis
Keywords: acute diarrhea; probiotics; children

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- probiotic (Placebo Comparator): Probiotic product with Sacharomices Boulardii
  Interventions: Drug: Placebo probiotic
- probiotic yogurt (Active Comparator): Yogurt with Lactobacilus Rhamnonsus strain spp
  Interventions: Dietary Supplement: Probiotic yogurt

INTERVENTIONS:
Dietary Supplement: Probiotic yogurt — Lactobacilus Rhamnonsus 100000000 UFC per mL. Dosage 50 mL twice daily fo 5 days.
  Arms: probiotic yogurt
Drug: Placebo probiotic — Lyophilized probiotic, containing 250 mg per sachet dosage to about 2 times a day for 5 days.
  Other Names: Florestor
  Arms: probiotic

SUMMARY:
The purpose of this study is to determine the effect of probiotic yogurt in acute watery diarrhea in children. The investigators will compare the effect of two different probiotics products.

DETAILED DESCRIPTION:
Background: Acute Gastroenteritis is one of the most and frequent disease in the childhood, considering the advances in treatment, Lactobacillus Rahmnosus has being well described as a probiotic who reduces the number of days of hospitalization and also de the severity.

Objectives: To evaluate the effect of the probiotic yogurt in the treatment of children who are between 10 months and 3 years old with acute non-dysenteric diarrhea.

Methods: A randomized clinical trial, controlled, double-blind. The investigators will have two groups of patients : One group will receive Lactobacillus Rahmnosus in a yogurt presentation and the other one will receive Sacharomyces boulardii in a lyophilized form ; the parameters of evaluation are going to be the number of diarrhea stools by day, number of vomiting episodes, hours with fever, nutritional and immunization state.

ELIGIBILITY:
Inclusion Criteria:

* All acute diarrhea

Exclusion Criteria:

* Severe malnourishment
* Severe dehydration
* Systemic infections

Ages: 10 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Duration of diarrhea | five days
  participants will be followed for the duration of hospital stay, an expected average of 5 days

SECONDARY OUTCOMES:
Duration of fever | five days
  participants will be followed for the duration of hospital stay, an expected average of 5 days
duration of vomiting | five days
  participants will be followed for the duration of hospital stay, an expected average of 5 days
duration of hospitalization | five days
  participants will be followed for the duration of hospital stay, an expected average of 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe E Grandy, MD MSc, Principal Investigator — Centro Pediatrico Albina Patino; Richard M Soria, MD, Study Director — Centro Pediatrico Albina Patino; Sdenka Jose, MD, Study Chair — Centro Pediatrico Albina Patino
Locations (1):
- Centro Pediatrico Albina Patino, Cochabamba, Departamento de Cochabamba, Bolivia